CLINICAL TRIAL: NCT04056000
Title: The Regulation of Fat Metabolism in a Cyclist With Lipodystrophy: a Case Study
Brief Title: Lipodystrophy and Fat Metabolism During Exercise
Acronym: FAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical and governance issues not resolved
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 258840
Record Dates: First submitted 2019-05-23; First posted 2019-08-14 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Healthy; Lipodystrophy, Familial Partial
MeSH Terms: conditions — Lipodystrophy, Familial Partial | interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercising following the ingestion of a high-carbohydrate br (Experimental): 60 minutes of cycling, with the ingestion of a high-carbohydrate breakfast and 200 mg of caffeine.
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: High-carbohdyrate breakfast; Behavioral: 60-minutes of steady state exercise
- Exercising following the ingestion of caffeine only (Experimental): 60 minutes of cycling, with the ingestion of 200 mg of caffeine.
  Interventions: Dietary Supplement: Caffeine; Behavioral: 60-minutes of steady state exercise
- Exercising in the absence of breakfast or caffeine ingestion (Experimental): 60 minutes of cycling, without the ingestion of breakfast, or caffeine.
  Interventions: Behavioral: 60-minutes of steady state exercise

INTERVENTIONS:
Dietary Supplement: Caffeine — 200 mg of caffeine, 60 minutes before exercise
  Arms: Exercising following the ingestion of a high-carbohydrate br; Exercising following the ingestion of caffeine only
Dietary Supplement: High-carbohdyrate breakfast — Ingestion of a high-carbohydrate breakfast 60 minutes before exercise
  Arms: Exercising following the ingestion of a high-carbohydrate br
Behavioral: 60-minutes of steady state exercise — See intervention name

SUMMARY:
Mandibular dysplasia with deafness and progeroid features (MDP) syndrome is a rare genetic metabolic disorder that causes lipodystrophy: the inability of the body to store subcutaneous adipose tissue (fat under the skin). This creates a unique scenario where any ingested fat is diverted to the abdomen and liver, often leading to diabetes.

The investigators have an opportunity to study an individual with MDP who has competed in and won national para-cycling championships and is able to prevent/control his diabetes by regular bicycle training. He has approached us for advice on nutritional strategies to improve his cycling performance, and insight into how he uses fat during exercise.

The investigators also wish to study a moderately-trained cyclist with Familial partial lipodystrophy (FPL). Those with FPL show a different pattern of lipodystrophy than those with MDP, allowing us to further increase the investigator's understanding of fat utilisation in those with lipodystrophy during exercise.

The investigators know how subcutaneous fat is used during exercise, and how duration, nutrition, carbohydrate availability, and exercise intensity can affect this. The investigators aim to investigate these processes during exercise in MDP and FPL. This will potentially provide nutrition and performance advice to the individuals, and insight on fat use in lipodystrophy and diabetes.

DETAILED DESCRIPTION:
During prolonged sub-maximal endurance exercise, both fat and carbohydrate are readily used substrates. The relative contribution and regulation of either is dependent on substrate availability (endogenous and exogenous), the duration of exercise, and the intensity of exercise. For example, exercising under fasted or caffeine supplemented conditions increases adipose tissue lipolysis, free fatty acid availability, and thus fat utilisation, whilst exercising under fed or carbohydrate loaded conditions increases glucose availability from elevated liver and muscle glycogen stores, and thus carbohydrate utilisation. This is important during prolonged sub-maximal exercise because when the limited endogenous carbohydrate stores are depleted, the body must rely more on fat. However, it is not known whether this regulation is present in conditions such as MDP and FPL where there is essentially no adipose tissue.

The investigators have an opportunity to study an individual with MDP who has competed in and won national para-cycling championships. He has approached us for advice on nutritional strategies to improve his cycling performance, and insight into how he uses fat during exercise. Intriguingly, the individual has provided anecdotal evidence that exercising under fasted conditions severely impairs his performance but that the use of caffeine improves his performance. He also states that he uses carbohydrate feeding strategies before and during prolonged exercise but is unsure whether it helps or not. This raises two fundamental questions that should be answered before any nutritional advice should be given (e.g. should a pre-exercise fat feeding or low glycemic index carbohydrate strategy be adopted?):

1. Do fasting and caffeine stimulate lipolysis in lipodystrophy and, if so, where is the fat coming from?
2. Does carbohydrate feeding before exercise impair lipolysis in lipodystrophy?

In order to answer these questions, the investigators need to directly measure rates of fat and carbohydrate utilisation from the circulation and muscle stores during exercise in the individual and a control participant using a stable isotope infusion approach. As well as providing results of significant scientific interest to the lipodystrophy field (researchers, clinicians, patients) and answering fundamental exercise physiology questions on substrate availability, the investigators hope that the outcomes will offer a substantial platform for improving the participant's knowledge of exercise nutrition and exercise performance.

ELIGIBILITY:
SUBJECT WITH FPL

Inclusion:

• Already known to researchers. Male, 29 years old.

CONTROL SUBJECT 1

Inclusion:

* Highly trained, elite-level cyclist (VO2max > 80 ml/kg/min)
* Registered with, and racing under the jurisdiction of, British Cycling
* ~< 10% of body fat
* Male
* 18 - 35 years old

Exclusion:

* Any diagnosed metabolic impairment, as this may affect normal metabolism.
* Any diagnosed cardiovascular disease or hypertension to avoid any complications associated with heavy exercise.
* Chronic use of any prescribed or over-the-counter pharmaceuticals.

CONTROL SUBJECT 2

Inclusion:

* Recreationally active, preferably with experience of cycling training.
* Similar (± 5 ml⋅kg-1⋅min-1) VO2max¬ to that of the participant with MDP

Exclusion:

* Any diagnosed metabolic impairment, as this may affect normal metabolism.
* Any diagnosed cardiovascular disease or hypertension to avoid any complications associated with heavy exercise.
* Chronic use of any prescribed or over-the-counter pharmaceuticals.

SUBJECT WITH FPL

Inclusion:

* Recreationally active, preferably with experience of cycling training.
* Similar (± 5 ml⋅kg-1⋅min-1) VO2max¬ to that of the participant with MDP
* Diagnosis with FPL

Exclusion:

* Female
* Any diagnosed cardiovascular disease or hypertension to avoid any complications associated with heavy exercise.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Substrate utilisation | Throughout the 60 minute cycle
  n..b. Please be aware that the below is a single, composite measure, wherein no single outcome measure cannot exist without the other. As such, it is presented as is, below.
  How carbohydrate and caffeine ingestion can affect the contribution to energy expenditure during 1 hour of exercise at 55%Wmax from:
  1. Plasma free fatty acids
  2. Plasma glucose
  3. Muscle glycogen
  4. Fat from other sources (predominantly muscle)
  This will be calculated from
  1. Plasma free fatty acid oxidation: Production of breath 13CO2 from a continuous infusion of [U-13C]palmitate
  2. Plasma glucose oxidation: The rate of disappearance of labelled [6, 6-2H2] glucose from a continuous infusion
  3. Muscle glycogen = Total carbohydrate oxidation - plasma glucose oxidation
  4. Fat from other sources = total fat oxidation - plasma free fatty acid oxidation

SECONDARY OUTCOMES:
Heart rate | Throughout the 60 minute cycle
  Heart rate will be measured throughout with the use of a heart rate monitor.
Plasma glucose concentrations | Throughout the 60 minute cycle
  A cannula will be used to draw blood from subjects at several time points. Whole blood samples will be analysed immediately for plasma glucose.
Plasma lactate concentrations | Throughout the 60 minute cycle
  A cannula will be used to draw blood from subjects at several time points. Whole blood samples will be analysed immediately for plasma lactate.
Plasma NEFA concentrations | Throughout the 60 minute cycle
  A cannula will be used to draw blood from subjects at several time points. At the end of the trial, plasma samples will be moved to a -80°C freezer for later analysis for NEFA.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davenport, MSc, Principal Investigator — The University of Exeter
Locations (1):
- School of Sport and Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No